CLINICAL TRIAL: NCT02195843
Title: Quadripolar Leads for the Management of Heart Failure Patients in the Middle East
Acronym: QUADRA-ME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Abdulmohsen Al Musa'ad, MD, Consultant Adult Cardiologist, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SA-2014-07-10
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Heart Failure
Keywords: CRT-D; Heart Failure; Middle East; Quadripolar
MeSH Terms: conditions — Heart Failure | interventions — Lead

ARMS (2):
- Emperical (Active Comparator): Anatomical optimization of device and leads
  Interventions: Other: Anatomical optimization of device and leads; Device: Implanted device and lead (Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and SJM Quadripolar lead system)
- Electrical (Active Comparator): Electrical optimization by RVLV Conduction Time with VectSelect
  Interventions: Other: Electrical optimization by RVLV Conduction Time with VectSelect; Device: Implanted device and lead (Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and SJM Quadripolar lead system)

INTERVENTIONS:
Other: Electrical optimization by RVLV Conduction Time with VectSelect — VectSelect Quartet multivector testing is a programmer-based feature that provides centralized vector testing and programming with the flexibility to select the appropriate pacing vector to meet individual patient needs.
  The Right ventricle - Left Ventricle (RV-LV) conduction time measurement will automatically identify the RV-LV conduction time for each LV electrode .
  Other Names: VectSelect Quartet multivector testing
  Arms: Electrical
Other: Anatomical optimization of device and leads — Patients will be implanted with left ventricular leads which will be positioned most basal, most apical or midway in the left ventricle. This follows the physician's routine clinical practice and judgement.
  Arms: Emperical
Device: Implanted device and lead (Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and SJM Quadripolar lead system) — All participants will be implanted with a St Jude Medical (SJM) Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and SJM Quadripolar lead system. Patients who fulfill the criteria for CRT D implant, will be invited to participate in this clinical investigation. Patients implanted with chronic leads requiring device upgrade to CRT-D can also be enrolled in the study, provided they are receiving a CRT-D device for the first time.

SUMMARY:
Heart failure is the most rapidly growing cardiovascular condition in developed countries. Despite advances in medical therapy, patients with heart failure are at high risk for death and hospitalization. Cardiac Resynchronization Therapy - defibrillators (CRT-D) are an effective treatment for heart failure.

Despite the high success rate of a CRT-D implant, there is a possibility of 10% that the LV lead cannot be implanted in patients undergoing a trans-venous system implantation. In this case, the patients may undergo multiple procedures before a lead is successfully implanted. These implant failures are not due to patient selection but rather to patients heart anatomy leading to lead stability problems, phrenic nerve stimulation (also called diaphragmatic stimulation) and poor electrical measurements.

The phrenic nerve is not part of the heart but runs near to this area on the way to a large muscle, called diaphragm, which separates the lung space from the space containing stomach, liver, kidneys and other internal organs in the abdomen. If the lead electrode is close to this nerve, it can cause a small part of it to contract giving you an uncomfortable hiccupping sensation.

In many patients, phrenic nerve stimulation is not identified until after the implant procedure when movement and postural changes bring the LV lead into closer contact with the phrenic nerve.

The investigation is performed to demonstrate the equality of performance of two different modalities of optimization of the implanted device and Quartet lead, Empirical (anatomical) optimization and Right Ventricle Left Ventricle (RVLV) conduction delay optimization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patient met standard CRT-D device indications (Left Ventricular Ejection Fraction (LVEF) ≤ 35%, QRS ≥ 120 ms, New York Heart Association (NYHA) Class II, III or ambulatory Class IV Heart Failure (HF) symptoms with optimal recommended medical therapy) and will be implanted with an St Jude Medical CRT-D
* Patient is willing to provide written informed consent.

Exclusion Criteria:

* Patient with non left bundle branch block (RBBB, intraventricular delay (IVCD) Block)
* Patient has an epicardial ventricular lead system.
* Patient has limited intrinsic atrial activity (≤ 40 bpm).
* Patient has persistent or permanent Atrial Fibrillation.
* Patient's life expectancy is less than 1 year
* Patient is pregnant.
* Patient is dependent on IV inotropic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular End Systolic Volume (LVESV) | 6 months post baseline
  Positive Clinical response defined as % change of Left Ventricular End Systolic Volume (LVESV) at 6 months follow up, compared to baseline